CLINICAL TRIAL: NCT05558033
Title: The Effects of Motor Imagery and Action Observation-Based Plyometric Training on Vastus Lateralis and Biceps Femoris Muscle Architectures of Adolescent Football Players
Brief Title: Motor Imagery and Muscle Architecture
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Murat EMİRZEOĞLU, Principal Investigator, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2022-11475
Record Dates: First submitted 2022-09-23; First posted 2022-09-28 (Actual); Last update posted 2022-11-29 (Actual); Status verified 2022-11

CONDITIONS: Muscle Architecture
Keywords: motor imagery; action observation; plyometric training; biceps femoris; vastus lateralis; muscle architecture; fiber length; pennation angle; muscle thickness; function; single leg jump
MeSH Terms: interventions — Plyometric Exercise

STUDY DESIGN:
Intervention Model Description: Parallel group randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Plyometric Training Group (Experimental): Individuals in the plyometric training group will receive plyometric training. In this training, individuals will not participate in a real plyometric training. Volunteers will watch videos to be prepared (action observation) and imagine them performing those exercises (motor imagery). All trainings will be given on the basis of telerehabilitation via distance education tools.
  Interventions: Other: Plyometric Exercise
- Control Group (Active Comparator): Athletes in this group will continue their routine training programs like the athletes in the plyometric training group.
  Interventions: Other: Football Training

INTERVENTIONS:
Other: Plyometric Exercise — Plyometric training consisting of ten different exercises [vertical unilateral and bilateral counter movement jump, horizontal unilateral and bilateral counter movement jump, drop jump (30 cm), squat jump, step-hop (20 cm), 180 degree rotation in transverse plane, frontal plane hurdle jump (20 cm) and sagittal plane hurdle jump (20 cm)] for 8 weeks, 3 sessions per week. Individuals will not participate in a real plyometric training. Volunteers will watch videos to be prepared (action observation) and imagine them performing those exercises (motor imagery)
  Arms: Plyometric Training Group
Other: Football Training — Routine football trainings
  Arms: Control Group

SUMMARY:
The aim of this study is to examine the effects of plyometric training on biceps femoris longus (BFl) and vastus lateralis (VL) muscle architecture in healthy football players. Individuals will be randomly placed into training and control groups. Measurements of muscle architecture will be taken bilaterally from BFl and VL muscles by means of an ultrasound device. Functional performance will be evaluated with the single leg jump test. Following the initial evaluations, individuals in the training group will receive plyometric training. Evaluations of muscle architecture and functional performance will be taken again from the individuals in the training and control groups at the end of the 4th and 8th weeks. The received ultrasound images will be calculated through the MicroDicom software. In-group and between-group comparisons will be analyzed using the Statistical Package for the Social Sciences program and appropriate tests.

DETAILED DESCRIPTION:
The aim of this study is to examine the effects of plyometric training on biceps femoris longus (BFl) and vastus lateralis (VL) muscle architecture (fiber length, penation angle and muscle thickness) in healthy football players. Individuals will be randomly placed into two different groups, the training group and the control group. Imagery ability, self-efficacy and motivation will be evaluated with various questionnaires and scales in order to compare the homogeneity of the groups. Measurements of muscle architecture will be taken bilaterally from BFl and VL muscles by means of an ultrasound device. Functional performance will be evaluated with the single leg jump test. Following the initial evaluations, individuals in the training group will receive plyometric training consisting of ten different exercises for 8 weeks, 3 sessions per week. In this training, individuals will not participate in a real plyometric training. Volunteers will watch videos to be prepared (action observation) and imagine them performing those exercises (motor imagery). All trainings will be given on the basis of telerehabilitation via distance education tools. Cognitive fatigue at the beginning and end of the session; at the end of each session, the technical quality and efficiency of the training will be evaluated. Evaluations of muscle architecture and functional performance will be taken again from the individuals in the control and training groups at the end of the 4th and 8th weeks. The received ultrasound images will be calculated through the MicroDicom software. In-group and between-group comparisons will be analyzed using the Statistical Package for the Social Sciences program and appropriate tests.

ELIGIBILITY:
Inclusion Criteria:

* Be in the 12-19 age range
* Being actively playing football as licensed

Exclusion Criteria:

* Those who have undergone lower extremity surgery
* Those with a history of second and third degree strain type injuries in the hamstring and quadriceps muscle groups
* Those with a history of injury to the lower extremity in the last two years
* Those with a history of congenital, neurological, orthopedic, rheumatological and cardiopulmonary pathologies or anomalies,
* Those with a diagnosis of systemic disease (diabetes, blood pressure, thyroid diseases, etc.)
* Those with acute infection and pain
* Those with a diagnosis of joint instability
* Those with a body mass index of 30 and above
* Those who received energy supplements or ergogenic aids during the study or during the 6-month period before the study
* Those who do not follow the research protocol

Ages: 12 Years to 19 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-11-21 (Actual); Primary Completion 2023-03-15 (Estimated); Study Completion 2023-06-15 (Estimated)

PRIMARY OUTCOMES:
Muscle Architecture Change-1 | Before, at the end of the fourth week and the eighth week
  Fiber length of the vastus lateralis and biceps femoris longus muscles
Muscle Architecture Change-2 | Before, at the end of the fourth week and the eighth week
  Pennation angle of the vastus lateralis and biceps femoris longus muscles
Muscle Architecture Change-3 | Before, at the end of the fourth week and the eighth week
  Muscle thickness of the vastus lateralis and biceps femoris longus muscles

SECONDARY OUTCOMES:
Functional Performance Change-1 | Before, at the end of the fourth week and the eighth week
  Single leg jump distance

CONTACTS AND LOCATIONS:
Overall Officials: Özlem Ülger, Study Director — Hacettepe University
Locations (1):
- Of Football Club, Trabzon, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided